CLINICAL TRIAL: NCT00781885
Title: A Multi-Center, Open-Label, Multiple Dose, Dose Finding Study Exploring the Safety and Tolerability of Beraprost Sodium Modified Release in PAH Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPS-MR-PAH-201
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Beraprost sodium modified release — Tablets 60mcg

SUMMARY:
This study is an international, open-label, multi-center, Phase II, multiple dose, dose-finding study to investigate the safety, tolerability and pharmacokinetic characteristics of BPS-MR tablets in male and female patients with PAH.

Patients who meet the inclusion/exclusion criteria will enter the Treatment Phase at a Baseline visit. Patients will begin taking one BPS-MR tablet (60µg) twice daily (b.i.d.) escalating by one tablet b.i.d. each week to a maximum dose of 600µg (ten tablets) b.i.d or until the patient reaches their MTD. Following the achievement of the MTD, patients will be down-titrated off BPS-MR in weekly one tablet b.i.d. decrements. Patients may, alternatively, elect to continue taking the study drug at their MTD in a separate open-label extension study.

DETAILED DESCRIPTION:
This study is an international, open-label, multi-center, Phase II, multiple dose, dose-finding study to investigate the safety, tolerability and pharmacokinetic characteristics of BPS-MR tablets in male and female patients with PAH. All patients will be receiving background therapy with either a phosphodiesterase (PDE-5) inhibitor, endothelin receptor antagonist (ERA), or the combination of these two.

The study is divided into two phases:

1. The Treatment Phase and
2. The Down-Titration Phase

Screening will be conducted on an outpatient basis within 21 days prior to the Baseline visit. Patients meeting the inclusion/exclusion criteria at the Baseline visit will enter the Treatment Phase and begin taking one BPS-MR tablet (60µg) b.i.d. and escalating by one tablet b.i.d. each week to a maximum dose of 600µg (ten tablets) b.i.d. or until the patient reaches an intolerable dose.

Patients who reach an intolerable dose will be instructed to continue treatment at the previous dose, which will be considered as their individual MTD. For example, if a patient attains a full week of six BPS-MR tablets b.i.d. (360µg) but is unable to tolerate seven tablets (420µg) then the patient will return to using six tablets of BPS-MR b.i.d. (360µg) for up to an additional week of treatment. In this scenario, BPS-MR 360µg b.i.d. is the patient's MTD. Patients who do not reach an intolerable dose and tolerate the full ten weeks of BPS-MR dosing will be considered to have their individual MTD as BPS-MR 600µg b.i.d.

When patients reach their individual MTD (either at 10 weeks or earlier) they will return to the site 3-7 days after for an End of Treatment Phase assessment to be evaluated for safety and, optionally, a PK assessment. Subsequent to the End of Treatment Phase visit patients will be instructed to begin down-titration off of BPS-MR in weekly increments. However, patients may alternatively elect to continue taking BPS-MR at their MTD in a separate open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female between the ages of 18 and 75 years of age, inclusive;
2. Has either idiopathic or familial PAH, PAH associated with collagen vascular disease, or PAH induced by anorexigens;
3. Is clinically stable, as determined by the investigator;
4. Has previously undergone a cardiac catheterization which is consistent with PAH, specifically PAPm ≥25 mmHg (at rest), PCWP (or left ventricular end diastolic pressure) ≤15 mmHg, and PVR >3 wood units;
5. Has been on a course of an endothelin receptor antagonist (ERA) or phosphodiesterase inhibitor (PDE-5) or the combination for at least 90 days at the time of the Baseline visit;
6. Has an unencouraged six-minute walk distance (6MWD) between 300 and 600 meters at the Screening visit;
7. Is able to communicate effectively with study personnel;
8. Is considered to be reliable, willing, cooperative and compliant with the study protocol requirements;
9. Provides voluntary, written informed consent before participating in the study;
10. Is, if female, physiologically incapable of childbearing or is practicing an acceptable method of birth control (i.e., surgical sterilization, approved hormonal contraceptives, barrier methods [such as a condom or diaphragm] used with a spermicide, or an intrauterine device).

Exclusion Criteria:

1. Has pulmonary venous hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis, severe chronic obstructive pulmonary disease, pulmonary hypertension related to congenital heart disease, or chronic thromboembolic pulmonary hypertension;
2. Is pregnant or lactating;
3. Has a known intolerance to beraprost sodium or prostanoids;
4. Has a pre-existing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs;
5. Current use of tobacco products;
6. Known history of syncope;
7. Has, in the opinion of the Investigator, any concomitant disease other than those accepted as part of the inclusion criteria that would compromise the patient or the study;
8. Has had a change in or discontinued any PAH medication (with the exception of anticoagulants) within 30 days prior to the Baseline visit;
9. Has received any prostanoid therapy within the 30 days prior to the Baseline visit or be scheduled to receive additional prostanoid therapy during the study except for acute vasodilatory testing;
10. Has received any investigational medication within 30 days prior to the Baseline visit or be scheduled to receive another investigational drug during the course of this study;
11. In the opinion of the investigator, may be unable to comply with the study protocol;
12. Has any preexisting disease known to cause pulmonary hypertension (e.g., obstructive lung disease, parasitic disease affecting the pulmonary system, sickle cell anemia, mitral valve stenosis, portal hypertension) other than those listed in the inclusion criteria;
13. Has donated blood or plasma or has lost a volume of blood >450 mL within six weeks prior to the Baseline visit.
14. Has an ongoing hemorrhagic condition (e.g. upper digestive track hemorrhage, hemoptysis, etc.) or has a pre-existing condition that, in the investigator's judgement, may increase the risk for developing hemorrhage during the study (e.g. hemophilia). However, transient hemorrhage (e.g. epistaxis, normal menstrual bleeding, gingival bleeding, hemorrhoidal hemorrhage, etc.) would not preclude enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01-31 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Staub, MS, MEng, Study Director — Study Sponsor
Locations (6):
- United States (3):
  - Harbor-UCLA Medical Center, Torrance, California
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UTSW Medical Center, Dallas, Texas
- Belgium (2):
  - Universite Libre de Bruxelles, Hospital Erasme, Brussels
  - Gastuiberg University Hospital, Leuven
- Mater Misericordiae University Hospital Ltd., Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Protocol Amendment was to include an optional arm investigating Beraprost Sodium Modified Release Tablets administered four times daily (QID), however, no participants were enrolled into this arm.
Groups:
- Beraprost Sodium: Beraprost Sodium Modified Release (BPS-MR) 60 mcg tablets, administered orally, twice daily (BID). Doses were escalated by 1 tablet BID weekly, as tolerated, to a maximum dose of 600 mcg BID.
Period: Overall Study
Arm/Group | Beraprost Sodium
Started | 19
Received at Least 1 Dose of Study Drug | 19
Completed | 18
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (7.57)
Respiratory Rate [Mean (Standard Deviation); unit: Breaths per minute] — Population: Only Participants with both a measurement at baseline and at the given visit are presented.
  Breaths per minute
    number analyzed (Participants) | 13
    (all) | 18.5 (1.61)
Temperature [Mean (Standard Deviation); unit: degrees Celsius] — Population: Only Participants with both a measurement at baseline and at the given visit are presented.
  degrees Celsius
    number analyzed (Participants) | 15
    (all) | 36.5 (0.35)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 118.1 (10.9)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 76.8 (9.14)
Weight [Mean (Standard Deviation); unit: kg] | 81.7 (20.79)
Electrocardiogram (ECG) Intervals [Mean (Standard Deviation); unit: msec] — Population: Only Participants with both a measurement at baseline and at the given visit are presented.
  msec
    PR Interval: number analyzed (Participants) | 18
    PR Interval | 175.8 (28.26)
    QRS Interval | 99.2 (14.7)
    QT Interval | 396.5 (42.1)
    QTc Bazett | 437.7 (27.4)
    QTc Friderica | 422.9 (28.65)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BPS-MR in Pulmonary Arterial Hypertension (PAH) Patients, Following Chronic, Twice-daily Administration.
Time Frame: 10 Weeks
Population: The Tolerability population includes all evaluable participants who achieved their MTD and had an End of Treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
Participants
  120 mcg | 2
  180 mcg | 2
  240 mcg | 3
  300 mcg | 2
  420 mcg | 1
  540 mcg | 1
  600 mcg | 7

2. Secondary Outcome: Number of Participants That Reported at Least One Treatment-Emergent Adverse Event (TEAE)
Description: A treatment-emergent adverse event (TEAE) is defined as an event not present prior to the initiation of the treatment or any event already present that worsens in either intensity or frequency following exposure to the treatment. AEs occurring more than 3 days after the last day study drug was taken in the study was not included in the statistical analyses or summaries (except for subjects with adverse events leading to study drug withdrawn). Only TEAEs that occurred during the treatment period of the BPS-MR-PAH-201 study were summarized. Any adverse event starting prior to the first dose of study drug was excluded from the summary analyses and only presented in the data listings. All efficacy results are descriptive; no statistical analysis was conducted
Time Frame: 19 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
Participants | 19

3. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline to Week 19
Description: Body Mass Index (BMI) was assessed at each study visit and taken after five minutes of seated rest. Body mass index is a value derived from the mass and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m², resulting from mass in kilograms and height in meters.
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: kilograms/meter^2
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
kilograms/meter^2 | -0.2 (0.98)

4. Secondary Outcome: Change in Weight From Baseline to Week 19
Description: Weight was assessed at each study visit and taken after five minutes of seated rest. Weight was measured in kilograms (kg).
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
kg | -0.5 (2.2)

5. Secondary Outcome: Change in Heart Rate From Baseline to Week 19
Description: Heart Rate was assessed at each study visit and taken after five minutes of seated rest. Heart rate is measured in beats per minute (BPM).
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: Beats per Minute (BPM)
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
Beats per Minute (BPM) | 0.7 (12.3)

6. Secondary Outcome: Change in Body Temperature From Baseline to Week 19
Description: Body Temperature was assessed at each study visit and taken after five minutes of seated rest. Body temperature was measured in degrees Celsius (C).
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
degrees Celsius | 0.1 (0.45)

7. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 19
Description: Systolic blood pressure was assessed at each study visit and taken after five minutes of seated rest. Systolic blood pressure was measured in millimeters of mercury (mmHg).
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
mmHg | 0.6 (12.46)

8. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Week 19
Description: Diastolic blood pressure was assessed at each study visit and taken after five minutes of seated rest. Diastolic blood pressure was measured in millimeters of mercury (mmHg).
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
mmHg | -2.5 (7.5)

9. Secondary Outcome: Change in Respiratory Rate From Baseline to Week 19
Description: Respiratory Rate was assessed at each study visit and taken after five minutes of seated rest. Respiratory rate was measured in breaths per minute.
Time Frame: Baseline and 19 weeks
Population: Participants with both a baseline measurement and an End of Study measurement
Measure: Mean (Standard Deviation); unit: Breaths per Minute
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
Breaths per Minute | 0.2 (1.24)

10. Secondary Outcome: Change in Electrocardiogram Intervals From Baseline to Week 19
Time Frame: Baseline and 19 weeks
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 19
millisecond (msec)
  PR Interval: number analyzed (Participants) | 18
  PR Interval | 6.1 (12.93)
  QRS Interval | -4.4 (12.46)
  QT Interval | 3.2 (29.37)
  QTc Bazett | -2.5 (20.05)
  QTc Friderica | -0.3 (21.59)

11. Secondary Outcome: Apparent Clearance (CL/F) of BPS-MR
Description: Apparent clearance is defined as plasma clearance divided by absolute bioavailability per kilogram of bodyweight.
Time Frame: pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 67
Population: 9 participants participated in the optional pharmacokinetic sub-study.
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 9
L/h/kg | 1.51 (0.52)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of BPS-MR
Time Frame: pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 67
Population: 9 participants participated in the optional pharmacokinetic sub-study.
Measure: Mean (Standard Deviation); unit: Liters per kilogram (L/kg)
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 9
Liters per kilogram (L/kg) | 43.6 (68.4)

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after study treatment discontinuation, up to 7 months.
Arm/Group | Beraprost Sodium
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beraprost Sodium (N=19)
Palpitations (Cardiac disorders) | 2
Cardiac Ventricular Disorder (Cardiac disorders) | 1
Ear Discomfort (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 6
Stomach Discomfort (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Defaecation Urgency (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Eye Injury (Injury, poisoning and procedural complications) | 1
Blood Bilirubin Increased (Investigations) | 1
Lymphocyte Count Increased (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Cold Sweat (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 7
Hot Flush (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days